CLINICAL TRIAL: NCT03576131
Title: First-in-human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety of GEN1029 in Patients With Malignant Solid Tumors
Brief Title: GEN1029 (HexaBody®-DR5/DR5) Safety Trial in Patients With Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1029-01; 2017-001394-16 (EudraCT Number); 236908 (Other: IRAS ID; UK Research Summaries Database)
Record Dates: First submitted 2018-05-08; First posted 2018-07-03 (Actual); Results first posted 2022-12-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Non-small Cell Lung Cancer; Triple Negative Breast Cancer; Renal Cell Carcinoma; Gastric Cancer; Pancreatic Cancer; Urothelial Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Carcinoma, Renal Cell; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1029 (HexaBody®-DR5/DR5) (Experimental)
  Interventions: Biological: GEN1029 (HexaBody®-DR5/DR5)

INTERVENTIONS:
Biological: GEN1029 (HexaBody®-DR5/DR5) — GEN1029 will be administered intravenously. The dose levels will be determined by the starting dose and the escalation steps taken in the trial.

SUMMARY:
The purpose of the trial is to evaluate the safety of GEN1029 (HexaBody®-DR5/DR5) in a mixed population of patients with specified solid tumors

DETAILED DESCRIPTION:
The trial is an open-label, multi-center first-in-human trial of GEN1029 (HexaBody®-DR5/DR5). The trial consists of two parts a dose escalation part (phase 1, first-in-human (FIH) and an expansion part (phase 2a). The expansion part of the trial will be initiated once the Recommended Phase 2 Dose (RP2D) has been determined.

ELIGIBILITY:
Inclusion Criteria (main):

* Patients with advanced and/or metastatic cancer who have no available standard therapy or who are not candidates for available standard therapy, and for whom, in the opinion of the investigator, experimental therapy with GEN1029 may be beneficial.
* Patient must be ≥ 18 years of age
* Patients must have measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
* Have an acceptable hematological status
* Have an acceptable renal function
* Have an acceptable liver function
* Have an Eastern Cooperative Oncology Group performance status of 0 or 1
* Body weight ≥ 40kg
* Patients both females and males, of childbearing or reproductive potential must agree to use adequate contraception from screening visit until six months after last infusion of GEN1029

Exclusion Criteria (main):

* Acute deep vein thrombosis or clinically relevant pulmonary embolism, not stable for at least 8 weeks prior to first GEN1029 administration
* Have clinically significant cardiac disease
* Have uncontrolled hypertension as defined in the protocol
* Any history of intracerebral arteriovenous malformation, cerebral aneurysm, new (younger than 6 months) or progressive brain metastases or stroke
* History of organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of Investigational Medicinal Product (IMP)
* Have received a cumulative dose of corticosteroid ≥ 150 mg prednisone (or equivalent doses of corticosteroids) within two weeks before the first GEN1029 administration
* History of ≥ grade 3 allergic reactions to monoclonal antibody therapy as well as known or suspected allergy or intolerance to any agent given in the course of this trial
* Radiotherapy within 14 days prior to first GEN1029 administration
* Any prior therapy with a compound targeting DR4 or DR5
* History of chronic liver disease or evidence of hepatic cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Plummer, Professor, Principal Investigator — Newcastle Hospitals NHS Foundation Trust
Locations (6):
- United States (2):
  - Yale University, New Haven, Connecticut
  - UT M.D Anderson Cancer Center, Houston, Texas
- Spain (2):
  - Hospital Univeritario Vall d'Hebron, Barcelona
  - START Madrid CIOCC, Madrid
- United Kingdom (2):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - The Royal Mardsen NHS Foundation Trust, Sutton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The sponsor decided to halt the development of GEN1029 due to a narrow therapeutic window after the dose-escalation part, hence the expansion part of the trial was not performed. Therefore, results are reported here only for the dose-escalation part.
Groups:
- Biweekly Regimen (GEN1029 0.1 mg/kg): Participants received 0.1 mg/kg of GEN1029 every 2 weeks (Q2W) until the end of treatment.
- Biweekly Regimen (GEN1029 0.2 mg/kg): Participants received 0.2 mg/kg of GEN1029 Q2W until the end of treatment.
- Biweekly Regimen (GEN1029 0.3 mg/kg): Participants received 0.3 mg/kg of GEN1029 Q2W until the end of treatment.
- Biweekly Regimen (GEN1029 1.0 mg/kg): Participants received 1.0 mg/kg of GEN1029 Q2W until the end of treatment.
- Biweekly Regimen (GEN1029 2.0 mg/kg): Participants received 2.0 mg/kg of GEN1029 Q2W until the end of treatment.
- Biweekly Regimen (GEN1029 3.0 mg/kg): Participants received 3.0 mg/kg of GEN1029 Q2W until the end of treatment.
- Priming Regimen (GEN1029 0.1 mg/kg): Participants received a priming dose of 0.1 mg/kg of GEN1029 on Cycle 1 Day 1. After 14 days and thereafter once every 14 days, participants received full dose of 0.3 mg/kg until the end of treatment.
- Intensified Regimen (GEN1029 1.0 mg/kg): Participants received 1.0 mg/kg of GEN1029 once a week (Q1W) for the first 8 weeks then Q2W until the end of treatment.
Period: Overall Study
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg) | Priming Regimen (GEN1029 0.1 mg/kg) | Intensified Regimen (GEN1029 1.0 mg/kg)
Started | 10 | 7 | 4 | 11 | 7 | 7 | 1 | 1
Completed | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 5 | 4 | 11 | 7 | 7 | 1 | 1
Not completed — Investigator decision | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 2 | 3 | 1 | 0
Not completed — Death | 3 | 3 | 1 | 5 | 4 | 1 | 0 | 1
Not completed — New anti-cancer treatment | 5 | 1 | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Unspecified reason | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Subject non-compliance | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least one dose of GEN1029 and were analyzed according to the actual trial treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg) | Priming Regimen (GEN1029 0.1 mg/kg) | Intensified Regimen (GEN1029 1.0 mg/kg) | Total
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7 | 1 | 1 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 2 | 7 | 3 | 4 | 1 | 0 | 27
  >=65 years | 3 | 4 | 2 | 4 | 4 | 3 | 0 | 1 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 2 | 8 | 5 | 4 | 1 | 0 | 27
  Male | 4 | 6 | 2 | 3 | 2 | 3 | 0 | 1 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 10 | 6 | 3 | 10 | 6 | 6 | 1 | 1 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  White | 8 | 5 | 3 | 11 | 7 | 7 | 1 | 1 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT criteria in the dose escalation phase of this trial are defined as hematologic toxicity including Grade (G) 4 neutropenia/thrombocytopenia for minimal duration of 7 days, G3/4 febrile neutropenia, >=G3 thrombocytopenia with bleeding, or G4 anemia; and non-hematologic toxicity including G4 infusion-related reactions (IRR) or anaphylaxis, G3 IRR did not resolve to =<G1 within 24 hours, >=G3 diarrhea/vomiting (did not respond to optimal treatment within 2 days), G3 nausea (did not respond to optimal treatment within 7days), or Hy's law or protocol-specified toxicities related to liver function test results or amylase and/or lipase elevations; or any >=G3 possibly related non-hematological AE, which occurred during first 2 cycles (as specified in protocol).
Time Frame: From Day 1 to 28 days after the first dose of study drug
Population: The Dose-Determining Set (DDS) consists of all participants from the Safety Set (received at least one dose of GEN1029 and analyzed according to the actual trial treatment received) who either received between 80% and 125% of the planned dose and completed the DLT observation period (Days 1-28), or experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 6 | 3 | 10 | 7 | 5
Participants | 0 | 1 | 0 | 3 | 3 | 2

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is defined as an AE that meets one of the following criteria: fatal or life-threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; medically significant (an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above [medical and scientific judgment must be exercised in deciding whether an AE is 'medically important']); required inpatient hospitalization or prolongation of existing hospitalization. A TEAE is defined as an AE occurring or worsening during the treatment period including the safety follow-up period.
Time Frame: Day 1 through Day 565 (corresponding to maximum observed duration)
Population: The Safety Set consists of all participants who received at least one dose of GEN1029 and analyzed according to the actual trial treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7
Participants
  Any TEAE | 8 | 7 | 4 | 11 | 7 | 7
  Any TESAE | 3 | 3 | 2 | 9 | 6 | 4

3. Primary Outcome: Number of Participants With >= Grade 3 Laboratory Results
Description: Number of participants with laboratory measurements of Grade >= 3 by NCI-CTCAE v4.03 are reported. The NCI-CTCAE is a descriptive terminology is used for AE reporting. The NCI-CTCAE v4.03 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE. Based on this general guideline: Grade 1 as mild AE, Grade 2 as moderate AE, Grade 3 as severe AE, Grade 4 as life-threatening or disabling AE, and Grade 5 as death. In case a participant reported multiple severity grades for an AE, only the maximum grade was used.
Time Frame: Day 1 through Day 565 (corresponding to maximum observed duration)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7
Participants
  Activated partial thromboplastin time prolonged | 0 | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 1 | 1 | 2 | 3 | 1 | 2
  Alkaline phosphatase increased | 0 | 0 | 1 | 0 | 1 | 0
  Amylase increased | 0 | 1 | 1 | 0 | 0 | 0
  Asparate aminotransferase increased | 1 | 2 | 0 | 0 | 0 | 2
  Bilirubin increased | 0 | 0 | 0 | 1 | 0 | 0
  Calcium decreased | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine increased | 1 | 0 | 0 | 0 | 0 | 0
  Gamma-glutamyl transferase increased | 2 | 2 | 1 | 2 | 3 | 1
  Glucose increased | 2 | 1 | 1 | 3 | 0 | 0
  Hemoglobin decreased | 0 | 1 | 0 | 0 | 0 | 0
  Lipase increased | 1 | 0 | 3 | 1 | 0 | 0
  Lymphocytes decreased | 2 | 3 | 1 | 2 | 2 | 0
  Magnesium increased | 0 | 0 | 0 | 0 | 0 | 1
  Prothrombin international normalized ratio - increased | 0 | 1 | 0 | 0 | 2 | 0
  Sodium decreased | 1 | 1 | 1 | 1 | 0 | 1
  Urate increased | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Hx-DR5-01 and Hx-DR5-05
Description: The Cmax of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: Pharmacokinetic (PK) analysis set included all participants who were exposed to at least 1 dose of GEN1029 and who had at least 1 post-dose PK measurement. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
µg/mL
  Cmax Hx-DR5-01 Cycle 1 (Day 1): number analyzed (Participants) | 9 | 6 | 4 | 11 | 7 | 6
  Cmax Hx-DR5-01 Cycle 1 (Day 1) | 0.86 (36.8) | 1.90 (38.0) | 2.81 (28.9) | 9.79 (20.9) | 21.31 (24.6) | 29.75 (24.9)
  Cmax Hx-DR5-01 Cycle 2 (Day 1): number analyzed (Participants) | 9 | 4 | 4 | 8 | 5 | 2
  Cmax Hx-DR5-01 Cycle 2 (Day 1) | 0.79 (42.9) | 2.11 (18.3) | 1.12 (59.9) | 8.36 (22.7) | 13.13 (156.3) | 29.56 (7.7)
  Cmax Hx-DR5-01 Cycle 3 (Day 1): number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 1
  Cmax Hx-DR5-01 Cycle 3 (Day 1) | 0.89 (16.6) | 1.82 (53.9) | 0.89 (146.4) | 7.20 (11.2) | 20.35 (24.7) | 28.80 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Cmax Hx-DR5-05 Cycle 1 (Day 1): number analyzed (Participants) | 9 | 6 | 4 | 11 | 7 | 6
  Cmax Hx-DR5-05 Cycle 1 (Day 1) | 0.87 (45.2) | 1.81 (35.7) | 2.82 (31.8) | 9.72 (17.0) | 20.90 (21.9) | 29.44 (27.9)
  Cmax Hx-DR5-05 Cycle 2 (Day 1): number analyzed (Participants) | 9 | 4 | 4 | 8 | 4 | 2
  Cmax Hx-DR5-05 Cycle 2 (Day 1) | 0.79 (25.9) | 2.00 (18.3) | 1.11 (76.2) | 7.75 (25.8) | 20.37 (14.3) | 30.52 (5.8)
  Cmax Hx-DR5-05 Cycle 3 (Day 1): number analyzed (Participants) | 7 | 4 | 2 | 6 | 3 | 1
  Cmax Hx-DR5-05 Cycle 3 (Day 1) | 0.87 (26.6) | 1.28 (93.8) | 1.62 (108.2) | 6.77 (20.6) | 5.27 (577.8) | 28.50 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

5. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to Infinity (AUC[0-inf]) of Hx-DR5-01 and Hx-DR5-05
Description: The AUC(0-inf) of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: PK analysis set included all participants who were exposed to at least 1 dose of GEN1029 and who had at least 1 post-dose PK measurement. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
µg*h/mL
  AUC(0-inf) Hx-DR5-01 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 7 | 6
  AUC(0-inf) Hx-DR5-01 Cycle 1 Day 1 | 39.44 (50.2) | 91.20 (66.0) | 85.80 (56.7) | 523.66 (47.5) | 1298.0 (22.7) | 1497.7 (58.7)
  AUC(0-inf) Hx-DR5-01 Cycle 2 Day 1: number analyzed (Participants) | 8 | 4 | 4 | 7 | 4 | 2
  AUC(0-inf) Hx-DR5-01 Cycle 2 Day 1 | 46.37 (61.5) | 105.32 (55.8) | 35.24 (30.5) | 530.48 (24.8) | 1071.5 (30.7) | 2488.5 (10.7)
  AUC(0-inf) Hx-DR5-01 Cycle 3 Day 1: number analyzed (Participants) | 6 | 4 | 2 | 6 | 3 | 1
  AUC(0-inf) Hx-DR5-01 Cycle 3 Day 1 | 37.43 (74.0) | 53.24 (133.3) | 41.41 (84.9) | 422.32 (26.8) | 1097.8 (36.6) | 2653.5 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  AUC(0-inf) Hx-DR5-05 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 6 | 6
  AUC(0-inf) Hx-DR5-05 Cycle 1 Day 1 | 32.97 (55.4) | 71.21 (66.9) | 83.37 (51.7) | 508.76 (33.0) | 1052.1 (24.7) | 1270.0 (60.1)
  AUC(0-inf) Hx-DR5-05 Cycle 2 Day 1: number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 2
  AUC(0-inf) Hx-DR5-05 Cycle 2 Day 1 | 39.31 (65.9) | 93.11 (66.6) | 44.76 (184.4) | 414.90 (24.1) | 609.90 (55.2) | 2273.6 (9.0)
  AUC(0-inf) Hx-DR5-05 Cycle 3 Day 1: number analyzed (Participants) | 5 | 3 | 2 | 6 | 2 | 1
  AUC(0-inf) Hx-DR5-05 Cycle 3 Day 1 | 25.87 (57.3) | 51.36 (161.6) | 67.23 (200.5) | 231.49 (53.2) | 412.87 (64.1) | 2398.5 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

6. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to the Time of Last Nonzero Concentration (AUC[0-Clast]) of Hx-DR5-01 and Hx-DR5-05
Description: The AUC(0-Clast) of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
µg*h/mL
  AUC(0-Clast) Hx-DR5-01 Cycle 1 Day 1: number analyzed (Participants) | 9 | 6 | 4 | 11 | 7 | 6
  AUC(0-Clast) Hx-DR5-01 Cycle 1 Day 1 | 24.36 (73.2) | 72.25 (70.6) | 60.78 (35.8) | 460.37 (43.5) | 1173.7 (15.6) | 1058.9 (88.6)
  AUC(0-Clast) Hx-DR5-01 Cycle 2 Day 1: number analyzed (Participants) | 9 | 4 | 4 | 8 | 5 | 2
  AUC(0-Clast) Hx-DR5-01 Cycle 2 Day 1 | 17.34 (141.3) | 70.33 (66.4) | 21.85 (36.0) | 308.74 (66.8) | 582.57 (84.8) | 2291.4 (18.1)
  AUC(0-Clast) Hx-DR5-01 Cycle 3 Day 1: number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 1
  AUC(0-Clast) Hx-DR5-01 Cycle 3 Day 1 | 22.34 (85.9) | 35.31 (151.4) | 6.85 (995.0) | 385.54 (23.7) | 986.38 (30.1) | 2444.7 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  AUC(0-Clast) Hx-DR5-05 Cycle 1 Day 1: number analyzed (Participants) | 9 | 6 | 4 | 11 | 7 | 6
  AUC(0-Clast) Hx-DR5-05 Cycle 1 Day 1 | 25.41 (120.7) | 53.76 (77.0) | 53.80 (50.8) | 432.18 (24.5) | 956.02 (18.8) | 964.48 (91.1)
  AUC(0-Clast) Hx-DR5-05 Cycle 2 Day 1: number analyzed (Participants) | 9 | 4 | 4 | 8 | 4 | 2
  AUC(0-Clast) Hx-DR5-05 Cycle 2 Day 1 | 24.85 (119.4) | 60.75 (76.0) | 29.17 (165.1) | 258.67 (60.5) | 395.50 (62.3) | 2176.0 (11.7)
  AUC(0-Clast) Hx-DR5-05 Cycle 3 Day 1: number analyzed (Participants) | 7 | 4 | 2 | 6 | 3 | 1
  AUC(0-Clast) Hx-DR5-05 Cycle 3 Day 1 | 20.12 (168.7) | 16.95 (539.4) | 43.56 (405.4) | 158.98 (76.4) | 52.16 (22162.5) | 2248.1 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

7. Secondary Outcome: Total Clearance (CL) of Hx-DR5-01 and Hx-DR5-05
Description: The CL of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
mL/h
  CL Hx-DR5-01 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 7 | 6
  CL Hx-DR5-01 Cycle 1 Day 1 | 95.98 (53.8) | 91.27 (51.4) | 123.75 (69.9) | 65.36 (56.5) | 59.07 (31.4) | 69.50 (51.0)
  CL Hx-DR5-01 Cycle 2 Day 1: number analyzed (Participants) | 8 | 4 | 4 | 7 | 4 | 2
  CL Hx-DR5-01 Cycle 2 Day 1 | 77.36 (70.2) | 79.97 (51.8) | 155.76 (72.6) | 58.07 (31.8) | 73.43 (28.0) | 36.92 (2.0)
  CL Hx-DR5-01 Cycle 3 Day 1: number analyzed (Participants) | 6 | 4 | 2 | 6 | 3 | 1
  CL Hx-DR5-01 Cycle 3 Day 1 | 99.53 (57.1) | 131.46 (76.0) | 111.33 (12.9) | 62.90 (42.5) | 62.64 (26.1) | 37.87 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  CL Hx-DR5-05 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 6 | 6
  CL Hx-DR5-05 Cycle 1 Day 1 | 111.10 (62.5) | 116.89 (51.3) | 127.35 (69.3) | 67.28 (37.4) | 69.39 (29.2) | 81.96 (53.9)
  CL Hx-DR5-05 Cycle 2 Day 1: number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 2
  CL Hx-DR5-05 Cycle 2 Day 1 | 90.18 (69.4) | 90.45 (67.1) | 131.51 (240.7) | 79.72 (28.8) | 134.11 (51.9) | 40.41 (3.7)
  CL Hx-DR5-05 Cycle 3 Day 1: number analyzed (Participants) | 5 | 3 | 2 | 6 | 2 | 1
  CL Hx-DR5-05 Cycle 3 Day 1 | 143.09 (50.5) | 140.38 (77.3) | 68.57 (42.2) | 114.74 (59.8) | 172.66 (78.9) | 41.90 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

8. Secondary Outcome: Volume of Distribution (Vss) at Steady State of Hx-DR5-01 and Hx-DR5-05
Description: The Vss of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
mL
  Vss Hx-DR5-01 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 7 | 6
  Vss Hx-DR5-01 Cycle 1 Day 1 | 5366.8 (35.0) | 4788.6 (5.0) | 3666.8 (49.4) | 3834.6 (34.3) | 4885.9 (18.8) | 4127.3 (19.2)
  Vss Hx-DR5-01 Cycle 2 Day 1: number analyzed (Participants) | 8 | 4 | 4 | 7 | 4 | 2
  Vss Hx-DR5-01 Cycle 2 Day 1 | 4720.0 (34.9) | 4287.5 (10.5) | 5283.0 (62.0) | 3998.1 (24.0) | 4185.8 (17.3) | 3427.5 (25.1)
  Vss Hx-DR5-01 Cycle 3 Day 1: number analyzed (Participants) | 6 | 4 | 2 | 6 | 3 | 1
  Vss Hx-DR5-01 Cycle 3 Day 1 | 4622.7 (31.1) | 4531.9 (6.7) | 3243.6 (14.3) | 4075.3 (26.2) | 4227.1 (8.7) | 4118.5 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Vss Hx-DR5-05 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 6 | 6
  Vss Hx-DR5-05 Cycle 1 Day 1 | 4722.7 (55.6) | 5242.9 (15.8) | 3942.4 (63.6) | 3611.0 (26.5) | 4291.6 (9.8) | 4142.9 (21.0)
  Vss Hx-DR5-05 Cycle 2 Day 1: number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 2
  Vss Hx-DR5-05 Cycle 2 Day 1 | 4899.3 (22.7) | 4701.6 (15.0) | 5177.9 (100.6) | 4054.4 (16.4) | 4334.9 (14.9) | 3187.8 (41.0)
  Vss Hx-DR5-05 Cycle 3 Day 1: number analyzed (Participants) | 5 | 3 | 2 | 6 | 2 | 1
  Vss Hx-DR5-05 Cycle 3 Day 1 | 4812.5 (31.9) | 5077.6 (24.1) | 3577.1 (15.7) | 4951.2 (42.4) | 5130.8 (5.6) | 4173.9 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

9. Secondary Outcome: Half-life Lambda-z (t1/2) of Hx-DR5-01 and Hx-DR5-05
Description: The t1/2 of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: as for outcome 5
Measure: Median (Full Range); unit: h
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
h
  T1/2 Hx-DR5-01 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 7 | 6
  T1/2 Hx-DR5-01 Cycle 1 Day 1 | 41.69 [20.7 to 61.1] | 41.31 [16.6 to 60.3] | 18.10 [11.4 to 40.5] | 40.27 [5.1 to 66.8] | 70.90 [50.5 to 86.2] | 42.45 [17.9 to 80.5]
  T1/2 Hx-DR5-01 Cycle 2 Day 1: number analyzed (Participants) | 8 | 4 | 4 | 7 | 4 | 2
  T1/2 Hx-DR5-01 Cycle 2 Day 1 | 37.75 [29.1 to 72.3] | 39.57 [21.7 to 62.5] | 24.47 [16.9 to 29.7] | 49.64 [36.2 to 71.5] | 33.62 [29.0 to 88.2] | 65.85 [54.6 to 77.1]
  T1/2 Hx-DR5-01 Cycle 3 Day 1: number analyzed (Participants) | 6 | 4 | 2 | 6 | 3 | 1
  T1/2 Hx-DR5-01 Cycle 3 Day 1 | 27.64 [16.2 to 84.1] | 19.93 [13.1 to 66.9] | 20.16 [16.2 to 24.1] | 47.86 [30.8 to 60.0] | 44.51 [40.1 to 64.0] | 77.00 [77.00 to 77.00]
  T1/2 Hx-DR5-05 Cycle 1 Day 1: number analyzed (Participants) | 8 | 6 | 4 | 11 | 6 | 6
  T1/2 Hx-DR5-05 Cycle 1 Day 1 | 35.55 [12.5 to 46.5] | 34.50 [15.6 to 52.5] | 19.10 [14.6 to 44.0] | 36.33 [26.4 to 70.6] | 42.68 [35.3 to 68.8] | 37.71 [16.6 to 69.6]
  T1/2 Hx-DR5-05 Cycle 2 Day 1: number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 2
  T1/2 Hx-DR5-05 Cycle 2 Day 1 | 32.46 [19.3 to 71.4] | 37.71 [17.3 to 80.7] | 25.43 [13.9 to 62.3] | 37.69 [28.4 to 43.5] | 26.68 [13.1 to 29.4] | 51.97 [30.8 to 73.1]
  T1/2 Hx-DR5-05 Cycle 3 Day 1: number analyzed (Participants) | 5 | 3 | 2 | 6 | 2 | 1
  T1/2 Hx-DR5-05 Cycle 3 Day 1 | 25.30 [12.0 to 39.6] | 18.75 [15.4 to 57.4] | 41.26 [24.3 to 58.2] | 33.90 [14.2 to 62.1] | 22.83 [13.2 to 32.5] | 70.9 [70.9 to 70.9]

10. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Hx-DR5-01 and Hx-DR5-05
Description: The Tmax of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: as for outcome 5
Measure: Median (Full Range); unit: h
Groups:
- 1. Biweekly Regimen (GEN1029 0.1 mg/kg): Participants received 0.1 mg/kg of GEN1029 every 2 weeks (Q2W) until the end of treatment.
- 2. Biweekly Regimen (GEN1029 0.2 mg/kg): Participants received 0.2 mg/kg of GEN1029 Q2W until the end of treatment.
- 3. Biweekly Regimen (GEN1029 0.3 mg/kg): Participants received 0.3 mg/kg of GEN1029 Q2W until the end of treatment.
- 4. Biweekly Regimen (GEN1029 1.0 mg/kg): Participants received 1.0 mg/kg of GEN1029 Q2W until the end of treatment.
- 5. Biweekly Regimen (GEN1029 2.0 mg/kg): Participants received 2.0 mg/kg of GEN1029 Q2W until the end of treatment.
- 6. Biweekly Regimen (GEN1029 3.0 mg/kg): Participants received 3.0 mg/kg of GEN1029 Q2W until the end of treatment.
Arm/Group | 1. Biweekly Regimen (GEN1029 0.1 mg/kg) | 2. Biweekly Regimen (GEN1029 0.2 mg/kg) | 3. Biweekly Regimen (GEN1029 0.3 mg/kg) | 4. Biweekly Regimen (GEN1029 1.0 mg/kg) | 5. Biweekly Regimen (GEN1029 2.0 mg/kg) | 6. Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
h
  Tmax Hx-DR5-01 Cycle 1 Day 1: number analyzed (Participants) | 9 | 6 | 4 | 11 | 7 | 6
  Tmax Hx-DR5-01 Cycle 1 Day 1 | 1.58 [1.1 to 5.8] | 1.89 [1.4 to 5.0] | 1.23 [1.2 to 1.4] | 2.00 [0.1 to 4.7] | 1.30 [1.1 to 3.6] | 1.46 [1.0 to 3.1]
  Tmax Hx-DR5-01 Cycle 2 Day 1: number analyzed (Participants) | 9 | 4 | 4 | 8 | 5 | 2
  Tmax Hx-DR5-01 Cycle 2 Day 1 | 1.25 [1.0 to 3.2] | 3.03 [3.0 to 5.2] | 1.30 [1.1 to 3.2] | 3.06 [1.1 to 5.1] | 3.25 [1.1 to 163.7] | 1.11 [1.0 to 1.2]
  Tmax Hx-DR5-01 Cycle 3 Day 1: number analyzed (Participants) | 7 | 4 | 3 | 6 | 3 | 1
  Tmax Hx-DR5-01 Cycle 3 Day 1 | 1.08 [0.0 to 3.4] | 1.48 [1.0 to 2.1] | 1.13 [1.1 to 1.3] | 3.08 [1.4 to 3.5] | 1.82 [1.1 to 3.2] | 3.1 [3.1 to 3.1]
  Tmax Hx-DR5-05 Cycle 1 Day 1: number analyzed (Participants) | 9 | 6 | 4 | 11 | 7 | 6
  Tmax Hx-DR5-05 Cycle 1 Day 1 | 1.75 [1.1 to 5.4] | 2.53 [1.0 to 4.8] | 2.36 [1.2 to 5.5] | 1.60 [0.1 to 4.7] | 1.35 [1.1 to 3.0] | 1.46 [1.0 to 3.1]
  Tmax Hx-DR5-05 Cycle 2 Day 1: number analyzed (Participants) | 9 | 4 | 4 | 8 | 4 | 2
  Tmax Hx-DR5-05 Cycle 2 Day 1 | 3.12 [1.1 to 5.1] | 2.19 [1.0 to 3.5] | 1.19 [1.0 to 1.4] | 2.26 [1.2 to 5.1] | 2.31 [1.1 to 3.3] | 2.21 [1.2 to 3.2]
  Tmax Hx-DR5-05 Cycle 3 Day 1: number analyzed (Participants) | 7 | 4 | 2 | 6 | 3 | 1
  Tmax Hx-DR5-05 Cycle 3 Day 1 | 1.08 [0.0 to 1.5] | 1.83 [1.0 to 3.3] | 1.18 [1.1 to 1.3] | 1.42 [1.1 to 3.0] | 1.13 [1.0 to 1.8] | 3.1 [3.1 to 3.1]

11. Secondary Outcome: Plasma Concentration of Hx-DR5-01 and Hx-DR5-05
Description: The plasma concentration of Hx-DR5-01 and Hx-DR5-05 are reported.
Time Frame: Predose, end of infusion, 2, 4, 24, 48, 168 and 336 hours after end of infusion on Day 1 of Cycles 1, 2, 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 11 | 7 | 6
µg/mL
  Plasma concentration Hx-DR5-01 Cycle 1 Day 1 (predose) | 0.085 (38.5) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0)
  Plasma concentration Hx-DR5-01 Cycle 2 Day 1 (predose): number analyzed (Participants) | 8 | 7 | 4 | 8 | 5 | 2
  Plasma concentration Hx-DR5-01 Cycle 2 Day 1 (predose) | 0.091 (61.0) | 0.075 (0.0) | 0.075 (0.0) | 0.084 (34.0) | 0.230 (77.8) | 0.283 (576.2)
  Plasma concentration Hx-DR5-01 Cycle 3 Day 1 (predose): number analyzed (Participants) | 7 | 5 | 3 | 6 | 3 | 1
  Plasma concentration Hx-DR5-01 Cycle 3 Day 1 (predose) | 0.075 (0.0) | 0.125 (164.3) | 0.075 (0.0) | 0.090 (46.4) | 0.224 (156.9) | 0.739 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Plasma concentration Hx-DR5-05 Cycle 1 Day 1 (predose) | 0.094 (77.6) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0)
  Plasma concentration Hx-DR5-05 Cycle 2 Day 1 (predose): number analyzed (Participants) | 8 | 7 | 4 | 8 | 5 | 2
  Plasma concentration Hx-DR5-05 Cycle 2 Day 1 (predose) | 0.097 (83.6) | 0.075 (0.0) | 0.075 (0.0) | 0.075 (0.0) | 0.155 (161.5) | 0.240 (372.5)
  Plasma concentration Hx-DR5-05 Cycle 3 Day 1 (predose): number analyzed (Participants) | 7 | 5 | 3 | 6 | 3 | 1
  Plasma concentration Hx-DR5-05 Cycle 3 Day 1 (predose) | 0.101 (94.6) | 0.119 (138.5) | 0.075 (0.0) | 0.094 (58.8) | 0.075 (0.0) | 0.568 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

12. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs) Positive to GEN1029
Description: From positive ADA samples titer values and neutralizing antibody scores (positive or negative) were determined and reported. A participant was considered positive if negative at baseline (screening) and had at least one positive post-baseline result, or positive at baseline and had at least one positive post-baseline result with a titer higher than baseline. Number of participants with ADA positive to GEN1029 are reported.
Time Frame: From Screening (Day -21 to -1) through Day 478 (corresponding to maximum observed duration)
Population: The Immunogenicity Set consists of all participants who received at least one dose of GEN1029 and analyzed according to the actual treatment received and had at least one immunogenicity measurement taken.
Measure: Count of Participants; unit: Participants
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7
Participants | 5 | 5 | 4 | 7 | 5 | 0

13. Secondary Outcome: Change From Baseline in Anti-tumor Activity Measured by Tumor Shrinkage
Description: Anti-tumor activity measured by tumor shrinkage was evaluated on based on of sum of the diameter(s) of all target lesions from the computerized tomography (CT) scan/positron emission tomography (PET)-CT scan. Largest tumor shrinkage is reported.
Time Frame: From Baseline (Day 1) through 8.8 months (corresponding to maximum observed duration)
Population: Full analysis set included all participants who received at least one dose of GEN1029 and were analyzed according to the actual treatment received.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 9 | 7 | 4 | 10 | 7 | 4
millimeter | 12.0 (11.843) | 12.0 (17.616) | 13.75 (9.032) | 1.10 (9.049) | 9.0 (10.909) | 15.50 (18.574)

14. Secondary Outcome: Number of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: The radiological evaluation was based on RECIST v1.1 using CT scan/PET-CT scan. The OR was defined as complete response (CR) or partial response (PR) per RECIST v1.1. The CR was defined as disappearance of all target and non-target lesions and reduction in short axis to <10 mm of any pathological and non-pathological lymph nodes. The PR was defined as >=30% decrease in sum of diameters of target lesions (compared to baseline), no unequivocal progression of existing non-target lesions, and no new lesion.
Time Frame: From Day 1 through 8.8 months (corresponding to maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST 1.1
Description: The PFS was defined as the number of days from the date of first study drug administration to first progressive disease (PD) or death from any cause. The PD was defined as at least 20% (and >= 5 mm) increase in the sum of the longest diameter (LD) of target lesions, compared to the smallest sum of the target LDs recorded while in trial or the appearance of 1 or more new lesions; unequivocal progression of existing non-target lesions; and/or new lesion. The radiological evaluation based on RECIST v1.1 was assessed using CT scan/PET scan. The PFS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 8.8 months (corresponding to maximum observed duration)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7
months | 2.5 [0.5 to 3.9] | 1.4 [0.5 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 2.4 [0.8 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 1.9 [1.2 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 1.2 [1.1 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 1.2 [1.0 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis.

16. Secondary Outcome: Overall Survival (OS) According to RECIST 1.1
Description: Overall survival was defined as the number of days from date of first study drug administration to death due to any cause. If a subject was not known to have died, then OS was censored, and the censoring date was the latest date the subject was known to be alive (on or before the cut-off date). The OS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 8.8 months (corresponding to maximum observed duration)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 10 | 7 | 4 | 11 | 7 | 7
months | 7.0 [2.3 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 6.4 [1.8 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 4.9 [NA to NA] — 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 7.1 [1.7 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 4.7 [2.8 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis. | 6.9 [NA to NA] — 95% confidence interval was not reached due to insufficient events being observed at the time of the analysis.

17. Secondary Outcome: Duration of Response (DoR) According to RECIST 1.1
Description: The radiological evaluation based on RECIST v1.1 was assessed using CT scan/PET-CT scan. The DoR was defined as duration from the first documentation of confirmed OR (CR or PR) to date of first progressive disease (PD) or death.
Time Frame: From Day 1 through 8.8 months (corresponding to maximum observed duration)
Population: Full analysis set included all participants who received at least one dose of GEN1029 and were analyzed according to the actual trial treatment received. Participants who achieved confirmed OR by the investigator assessment were evaluated for this outcome measure.
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Time to Response (TTR) According to RECIST 1.1
Description: TTR is defined as the number of days from first dose of study drug to the first documented confirmed CR or PR, which must be subsequently confirmed.
Time Frame: From Day 1 through 8.8 months (corresponding to maximum observed duration)
Population: as for outcome 17
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For AEs: Day 1 through Day 565 (corresponding to maximum observed duration); and for All-cause mortality: From date of informed consent through Day 565 (corresponding to maximum observed duration)
Arm/Group | Biweekly Regimen (GEN1029 0.1 mg/kg) | Biweekly Regimen (GEN1029 0.2 mg/kg) | Biweekly Regimen (GEN1029 0.3 mg/kg) | Biweekly Regimen (GEN1029 1.0 mg/kg) | Biweekly Regimen (GEN1029 2.0 mg/kg) | Biweekly Regimen (GEN1029 3.0 mg/kg) | Priming Regimen (GEN1029 0.1 mg/kg) | Intensified Regimen (GEN1029 1.0 mg/kg)
All-Cause Mortality (participants affected / at risk) | 3/10 | 3/7 | 1/4 | 5/11 | 4/7 | 1/7 | 0/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/10 | 3/7 | 2/4 | 9/11 | 6/7 | 4/7 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 8/10 | 7/7 | 4/4 | 11/11 | 7/7 | 7/7 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biweekly Regimen (GEN1029 0.1 mg/kg) (N=10) | Biweekly Regimen (GEN1029 0.2 mg/kg) (N=7) | Biweekly Regimen (GEN1029 0.3 mg/kg) (N=4) | Biweekly Regimen (GEN1029 1.0 mg/kg) (N=11) | Biweekly Regimen (GEN1029 2.0 mg/kg) (N=7) | Biweekly Regimen (GEN1029 3.0 mg/kg) (N=7) | Priming Regimen (GEN1029 0.1 mg/kg) (N=1) | Intensified Regimen (GEN1029 1.0 mg/kg) (N=1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea Versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prothrombin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biweekly Regimen (GEN1029 0.1 mg/kg) (N=10) | Biweekly Regimen (GEN1029 0.2 mg/kg) (N=7) | Biweekly Regimen (GEN1029 0.3 mg/kg) (N=4) | Biweekly Regimen (GEN1029 1.0 mg/kg) (N=11) | Biweekly Regimen (GEN1029 2.0 mg/kg) (N=7) | Biweekly Regimen (GEN1029 3.0 mg/kg) (N=7) | Priming Regimen (GEN1029 0.1 mg/kg) (N=1) | Intensified Regimen (GEN1029 1.0 mg/kg) (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (3) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 3 (3) | 4 (6) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 2 (5) | 2 (3) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (8) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 3 (5) | 2 (5) | 6 (14) | 3 (3) | 2 (2) | 1 (2) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 4 (6) | 2 (5) | 7 (14) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spider vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Results of the biweekly dosing regimens are based on the Clinical Study Report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 12 months but less than 18 months from the end of study (database lock).The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT03576131/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03576131/SAP_001.pdf